CLINICAL TRIAL: NCT07227779
Title: A PHASE 2 NOVEL ANTIMICROBIAL COMBINATION THERAPY TO TREAT TUBERCULOUS MENINGITIS
Brief Title: B-PaLMZ for TB Meningitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Infectious Diseases Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00024610
Record Dates: First submitted 2025-11-11; First posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Tuberculous Meningitis
MeSH Terms: conditions — Tuberculosis, Meningeal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BPaLMZ Regimen (Experimental): bedaquiline, pretomanid, linezolid, moxifloxacin, and pyrazinamide (BPaLMZ)
  Interventions: Drug: BPaLMZ Regimen
- Standard of Care Regimen (No Intervention): rifampicin, isoniazid, pyrazinamide, ethambutol (RHZE) therapy

INTERVENTIONS:
Drug: BPaLMZ Regimen — bedaquiline, pretomanid, linezolid, moxifloxacin, and pyrazinamide
  Arms: BPaLMZ Regimen

SUMMARY:
This two-stage study will compare consented research participants with tuberculous meningitis receiving BPaLMZ to controls receiving SOC of rifampicin (R), isoniazid (H), pyrazinamide (Z), and ethambutol (E), known as RHZE.

ELIGIBILITY:
Inclusion Criteria:

* First Episode definite or probable TBM with physician intent to treat
* Age ≥18 years
* Provision of Informed Consent by participant or surrogate
* Living with HIV
* Weight > 35kg, estimate or measured

Exclusion Criteria:

* Additional active and confirmed CNS infection
* Known rifampicin-resistant TB
* Allergy or contraindication to a study medicine
* More than 5 doses of any TB therapy received within the previous 14 days
* Presence of jaundice, known liver cirrhosis, elevated ALT or AST >3x ULN, or total bilirubin >2x ULN
* Estimated Glomerular Filtration Rate <30 ml/min/1.73m2
* Significant cardiac comorbidity, heart failure, arrhythmia, or QTc >450 ms
* Pregnancy or Breastfeeding
* Cryptococcal antigen positivity in blood
* Condition which makes participation not in the participant's best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to Death | 24 Weeks
Functional Status | 24 Weeks
  Modified Rankin score

CONTACTS AND LOCATIONS:
Overall Officials: David Boulware, MD, Principal Investigator — University of Minnesota
Locations (2):
- University of Minnesota, Minneapolis, Minnesota, United States
- Infectious Diseases Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes